CLINICAL TRIAL: NCT00709748
Title: The E-STIM Trial: A Randomized, Double-Blind, Multicenter Trial Comparing the Efficacy of the Empi Select Transcutaneous Electrical Nerve Stimulation (TENS) to a Control for the Treatment of Chronic Lower Back Pain
Brief Title: E-STIM Trial: Comparing the Efficacy of the Empi Select TENS to a Control for the Treatment of Chronic Lower Back Pain
Acronym: E-STIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Empi, A DJO Company (Industry)
Collaborators: Alquest (Industry)
Responsible Party: Jim Pomonis, PhD / Director of Clinical Programs, Empi, A DJO company
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Empi 07-1-02
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Lower Back Pain
Keywords: Transcutaneous electrical nerve stimulation; TENS; Empi; Electrotherapy; Back pain; Lower back pain; Chronic lower back pain
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects in this study arm will receive treatment (fully active) Empi Select TENS devices.
  Interventions: Device: Empi Select TENS Device
- 2 (Placebo Comparator): Subjects in this study arm will receive control (not fully active) Empi Select TENS devices.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Empi Select TENS Device — The Empi Select TENS device delivers therapeutic electrical currents at various frequencies (intensities) and periods of time for the treatment of pain.
  Other Names: -Transcutaneous electrical nerve stimulation; -TENS
  Arms: 1
Device: Placebo — Subjects in this study arm will receive control (not fully active) Empi Select TENS devices.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether transcutaneous electrical nerve stimulation (TENS) delivered via the Empi Select TENS device provides relief of chronic lower back pain.

DETAILED DESCRIPTION:
The E-STIM Trial is designed to collect data on the efficacy of the Empi Select Transcutaneous Electrical Nerve Stimulation (TENS) device for the treatment of chronic low back pain. This clinical trial is a non-significant risk, randomized, double-blinded, placebo-controlled 12-week trial involving the commercially available Empi Select TENS device for treating subjects with chronic (>90 days) low back pain. Multiple centers located in the United States will enroll approximately 300 subjects in this study. Eligible subjects will be randomized 1:1 to either the treatment group or the placebo group. The subjects and investigational staff are blinded to the treatment assignment. Subjects will return to the investigational center for follow-up assessments at 1, 4, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18-65 years of age.
* Subjects must have reported low back pain of at least 3 months duration.
* Subjects must report a low back pain score of 4 or greater on the 0-10 point Numerical Rating Scale (NRS) for average daily pain.
* Subjects must have been on a stabilized analgesic medication regimen for 3 months or greater.
* Subjects must be willing to discontinue use of all rescue pain medications for the duration of the trial (all PRN medications for breakthrough pain), except for OTC oral acetaminophen (up to 4 grams per day).
* Subjects must be willing to refrain from starting any new lower back pain treatments for the duration of the trial.
* Subjects must be willing and able to comply with all follow-up procedures (including completion of the daily diary) and return for scheduled follow- up visits.
* Female subjects must be post-menopausal for at least 1 year, surgically sterile or willing to take a pregnancy test which must be negative prior to study enrollment.
* Subjects must be willing and able to provide written informed consent and HIPAA authorization prior to enrollment into the study.

Exclusion Criteria:

* Subjects that have a demand type pacemaker or defibrillator.
* Subjects that have had previous experience with electrotherapy.
* Subjects that have had any failed back surgeries.
* Subjects that have spinal stenosis which contributes to, or is the cause of lower back pain.
* Subjects that have sciatica (lower back pain with radicular symptoms).
* Subjects that have cauda equina syndrome.
* Subjects that have fibromyalgia.
* Subjects that have pain secondary to cancer.
* Subjects who have cancer in the same anatomical location as their back pain.
* Subjects that have any sensory deprivation or diagnosis of shingles or post- herpetic neuralgia (specifically in the mid-trunk region).
* Subjects that have planned surgeries during the study period.
* Subjects that have a history of alcohol or substance abuse in the last 5 years.
* Subjects on psychoactive medication(s) that:

  1. have had a change in dose or a change in medication type during the 3 months prior to screening, or
  2. are expected to require a change in dose, or a new medication during the study.
* Subjects that are seeking worker's compensation or any other legal claims.
* Subjects that are pregnant or plan to become pregnant during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Relief of lower back pain as measured by a Numerical Rating Scale (NRS) of Average Daily Pain. | Baseline and at 1, 4, 8 and 12 week follow-up

SECONDARY OUTCOMES:
Improvement of function as measured by the Roland and Morris Back Pain Disability Scale. | Baseline and 1, 4, 8 and 12 week follow-up
Improvement of quality of life as measured by the SF-12 Health Survey. | Baseline and 1, 4, 8 and 12 week follow-up
Subject satisfaction as measured by the Patient Global Impression of Change scale (PGIC). | 1, 4, 8 and 12 week follow-up
Adverse Event Assessment: assess the occurrence and severity of any adverse events. | 1, 4, 8 and 12 week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jim Pomonis, PhD, Study Director — Empi, A DJO Company
Locations (8):
- United States (8):
  - MedInvestigations, Fair Oaks, California
  - Pain Consultants of West Florida, Pensacola, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Center for Prospective Outcome Studies, Atlanta, Georgia
  - Taylor Research LLC, Marietta, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Spinal Research Foundation, Reston, Virginia

REFERENCES:
- [Background] Johnson M, Martinson M. Efficacy of electrical nerve stimulation for chronic musculoskeletal pain: a meta-analysis of randomized controlled trials. Pain. 2007 Jul;130(1-2):157-65. doi: 10.1016/j.pain.2007.02.007. Epub 2007 Mar 23. PMID 17383095
- [Background] Deyo RA, Walsh NE, Martin DC, Schoenfeld LS, Ramamurthy S. A controlled trial of transcutaneous electrical nerve stimulation (TENS) and exercise for chronic low back pain. N Engl J Med. 1990 Jun 7;322(23):1627-34. doi: 10.1056/NEJM199006073222303. PMID 2140432
- [Background] Hamza MA, White PF, Ahmed HE, Ghoname EA. Effect of the frequency of transcutaneous electrical nerve stimulation on the postoperative opioid analgesic requirement and recovery profile. Anesthesiology. 1999 Nov;91(5):1232-8. doi: 10.1097/00000542-199911000-00012. PMID 10551571
- [Background] Graff-Radford SB, Reeves JL, Baker RL, Chiu D. Effects of transcutaneous electrical nerve stimulation on myofascial pain and trigger point sensitivity. Pain. 1989 Apr;37(1):1-5. doi: 10.1016/0304-3959(89)90146-2. PMID 2786179
- [Background] Cheing GL, Hui-Chan CW. Transcutaneous electrical nerve stimulation: nonparallel antinociceptive effects on chronic clinical pain and acute experimental pain. Arch Phys Med Rehabil. 1999 Mar;80(3):305-12. doi: 10.1016/s0003-9993(99)90142-9. PMID 10084439
- [Background] Sluka KA, Deacon M, Stibal A, Strissel S, Terpstra A. Spinal blockade of opioid receptors prevents the analgesia produced by TENS in arthritic rats. J Pharmacol Exp Ther. 1999 May;289(2):840-6. PMID 10215661
- [Background] Han JS, Chen XH, Sun SL, Xu XJ, Yuan Y, Yan SC, Hao JX, Terenius L. Effect of low- and high-frequency TENS on Met-enkephalin-Arg-Phe and dynorphin A immunoreactivity in human lumbar CSF. Pain. 1991 Dec;47(3):295-298. doi: 10.1016/0304-3959(91)90218-M. PMID 1686080
- [Background] Lee KH, Chung JM, Willis WD Jr. Inhibition of primate spinothalamic tract cells by TENS. J Neurosurg. 1985 Feb;62(2):276-87. doi: 10.3171/jns.1985.62.2.0276. PMID 3871474
- [Background] Garrison DW, Foreman RD. Effects of transcutaneous electrical nerve stimulation (TENS) on spontaneous and noxiously evoked dorsal horn cell activity in cats with transected spinal cords. Neurosci Lett. 1996 Sep 27;216(2):125-8. doi: 10.1016/0304-3940(96)13023-8. PMID 8904799
- [Background] Garrison DW, Foreman RD. Decreased activity of spontaneous and noxiously evoked dorsal horn cells during transcutaneous electrical nerve stimulation (TENS). Pain. 1994 Sep;58(3):309-315. doi: 10.1016/0304-3959(94)90124-4. PMID 7838579
- [Background] Khadilkar A, Milne S, Brosseau L, Wells G, Tugwell P, Robinson V, Shea B, Saginur M. Transcutaneous electrical nerve stimulation for the treatment of chronic low back pain: a systematic review. Spine (Phila Pa 1976). 2005 Dec 1;30(23):2657-66. doi: 10.1097/01.brs.0000188189.21202.0f. PMID 16319752
- [Background] Brosseau L, Milne S, Robinson V, Marchand S, Shea B, Wells G, Tugwell P. Efficacy of the transcutaneous electrical nerve stimulation for the treatment of chronic low back pain: a meta-analysis. Spine (Phila Pa 1976). 2002 Mar 15;27(6):596-603. doi: 10.1097/00007632-200203150-00007. PMID 11884907
- [Background] Ordog GJ. Transcutaneous electrical nerve stimulation versus oral analgesic: a randomized double-blind controlled study in acute traumatic pain. Am J Emerg Med. 1987 Jan;5(1):6-10. doi: 10.1016/0735-6757(87)90281-6. PMID 3545246